CLINICAL TRIAL: NCT01368263
Title: A Multisite International Collaborative Phase 2 Study of Neoadjuvant Goserelin and a Non-steroidal Aromatase Inhibitor for Premenopausal Women With Estrogen Receptor Positive HER2 Negative Clinical Stage 2 and 3 Breast Cancer
Brief Title: Goserelin and Letrozole or Anastrozole in Premenopausal Patients With Stage II-III Estrogen Receptor-Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to funding source and lack of accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201106141
Record Dates: First submitted 2011-06-02; First posted 2011-06-07 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Letrozole; Anastrozole; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Ki67 <10%, E2 <= 15 pg/ml) (Experimental): Patients receive 1 cycle (28 days) of endocrine therapy consisting of goserelin acetate SC on day 1 and letrozole or anastrozole PO QD. Neoadjuvant treatment repeats every 28 days for a total of 16-18 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo the appropriate standard surgical procedure to remove the cancer. Recommendations for postsurgical treatment will be based on PEPI score and physician discretion.
  Interventions: Drug: goserelin acetate; Drug: letrozole; Drug: anastrozole; Procedure: Surgery
- Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) (Experimental): Patients receive 1 cycle (28 days) of endocrine therapy consisting of goserelin acetate SC on day 1 and letrozole or anastrozole PO QD. Patients receive standard neoadjuvant chemotherapy in the absence of disease progression or unacceptable toxicity. Patients then undergo the appropriate standard surgical procedure to remove the cancer. Postsurgical treatment at physician discretion.
  Interventions: Drug: goserelin acetate; Drug: letrozole; Drug: anastrozole; Drug: chemotherapy; Procedure: Surgery
- Group 3 (E2 > 15 pg/ml) (Experimental): Patients receive 1 cycle (28 days) of endocrine therapy consisting of goserelin acetate SC on day 1 and letrozole or anastrozole PO QD. Patients receive standard neoadjuvant therapy at the discretion of the physician. Patients then undergo the appropriate standard surgical procedure to remove the cancer. Postsurgical treatment at physician discretion.
  Interventions: Drug: goserelin acetate; Drug: letrozole; Drug: anastrozole; Drug: chemotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: goserelin acetate — Given SC
  Other Names: ICI-118630; ZDX; Zoladex
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Drug: anastrozole — Given PO
  Other Names: ANAS; Arimidex; ICI-D1033
Drug: chemotherapy — Standard chemotherapy
  Other Names: chemo
  Arms: Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml); Group 3 (E2 > 15 pg/ml)
Procedure: Surgery

SUMMARY:
This phase II trial studies the impact of a presurgical endocrine therapy, consisting of goserelin with letrozole or anastrozole on the treatment of premenopausal patients with stage II-III estrogen receptor-positive (ER+) and human epidermal growth factor receptor 2 (HER2)-negative breast cancer. Endocrine therapy reduces the amount of estrogen in the body. E+ breast cancer require estrogen, so lower levels of estrogen may slow or stop cell growth. Giving goserelin together with letrozole or anastrozole before surgery may enhance the effectiveness of, or eliminate the need for, chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histological or cytological confirmed invasive breast cancer
* Patient must be premenopausal confirmed by serum estradiol level in the premenopausal range (> 25 pg/ml) at the beginning of the study; for women on oral contraceptives, these agents must be held for two weeks before the estradiol assessment is made
* Patient must have a negative serum pregnancy test within 7 days of registration
* Patient's tumor must be ER+ with or without concomitant progesterone receptor-positive (PR+) with an Allred score of 6, 7 or 8; patients with > 66.6% of cells staining positive by conventional immunohistochemistry (IHC) have a minimum Allred score of 6 and are eligible
* Patient's tumors must be HER2 negative by local laboratory assessment: HER2 IHC 0, 1+, or 2+ with subsequent negative fluorescent in situ hybridization (FISH) (ratio < 1.8); negative FISH alone in absence of IHC is acceptable
* Patient must have T2-T4c, any N, M0 breast cancer, by clinical staging (physical examination)
* Patient's primary tumor must be palpable and measure > 2 cm by tape, ruler or caliper measurements in at least one dimension
* Patient must have mammogram and ultrasound of the breast within 42 days prior to registration; if a patient has clinically palpable or suspicious nodes, then an ultrasound of the axilla is also required
* Patient, as documented by the treating physician, must be clinically staged as one of the following:

  * T4 a-c for which modified radical mastectomy with negative margins is the goal
  * T2 or T3 for which conversion from needing mastectomy to breast conservation is the goal
  * T2 for which lumpectomy at first attempt is the goal
* Patient must be > or = 18 years old.
* Patient must stop taking all forms of hormonal treatment, including oral or other form of hormonal contraceptive methods and all forms of hormone replacement therapy, at least two weeks prior to starting protocol therapy
* Patient must agree to use a "highly-effective form of non-hormonal contraception" (applies to patient and/or partner)
* Patient must be willing to undergo oophorectomy, if indicated
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patient must have normal organ and marrow function as defined below:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3.0 X institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* If the patient is a cancer survivor, all of the following criteria must be met
* Patient has undergone potentially curative therapy from all prior malignancies
* Patient must have no evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for successfully treated cervical carcinoma in situ, lobular carcinoma in situ of the breast, contralateral ductal carcinoma in situ (DCIS) treated with mastectomy or lumpectomy and radiation but without tamoxifen treatment, or non-melanoma skin cancer with no evidence of recurrence)
* Patient must be deemed by her treating physician to be at low risk (< 30%) for recurrence from prior malignancies
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patient must not have inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema)
* Patient must not have had prior treatment for invasive breast cancer, including radiation, endocrine therapy, chemotherapy, or investigational agent; patients whose diagnosis was established by incision biopsy are not eligible
* Patient must not have had prior DCIS in the ipsilateral breast
* Patient must not have used tamoxifen for prior contralateral DCIS
* Patient must not have any evidence of distant metastasis (M1) on imaging; staging scans are not mandatory but any exams performed as standard of care throughout the study period will be collected for correlation as needed
* If patient does not agree to undergo mastectomy or lumpectomy after neoadjuvant therapy, she is ineligible for this study
* Patient must not be receiving other investigational agents or be enrolled in another neoadjuvant clinical trial for treatment of the existing breast cancer
* Pregnant and/or breastfeeding women are excluded from this study
* Patient must not have any concurrent life threatening illnesses
* Patient must not have undergone prior sentinel lymph node surgery; cores or FNA of lymph node are acceptable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pluard, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant accrual on 09/13/2011 and closed to participant accrual on 05/22/2013.
Period: Overall Study
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Started | 6 | 1 | 1
Completed | 6 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml) | Total
Number analyzed (Participants) | 6 | 1 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] | 43 [35 to 53] | 29 [29 to 29] | 35 [35 to 35] | 38.5 [29 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 1 | 8
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (CR) Rate
Description: * In patients with Ki67 >10% and <= 15 pg/ml at 4 weeks.
  * The pCR rate for neo-adjuvant chemotherapy is defined as 100 times the number of eligible patients with no histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary or sentinel lymph nodes divided by the total number of eligible patients who received neo-adjuvant chemotherapy.
Time Frame: 1 month
Population: There were no evaluable participants to analyze in Group 1, 2, or 3. No participants met the criteria for Ki67 >10% and estradiol levels of <= 15 pg/ml at 4 weeks.
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Acceptability of Management With Surgical Oophorectomy/Continued LHRH With Continued Oral Endocrine Therapy and no Chemotherapy
Description: Proportion of patients with a PEPI score of 0 and pathological stage 1 who choose to forego chemotherapy.
Time Frame: 6 months post neoadjuvant endocrine therapy and surgery
Population: None of the participants had a PEPI score and 0 and pathological stage 1.
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Relationship Between Pretreatment FFNP-PET Standard Uptake Value (SUV) and 4-week Post-treatment Ki-67
Time Frame: Baseline and 4 weeks post-treatment
Population: This outcome was not analyzed due to funding issues.
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Preoperative Endocrine Prognostic Index Score (PEPI Score)
Description: To obtain the PEPI score, risk points for relapse-free survival (RFS) and breast cancer-specific survival (BCSS) are assigned depending on the hazard ratio (HR) from the multivariable analysis. The total PEPI score assigned to each patient is the sum of the risk points derived from the pT stage, pN stage, Ki67 level, and estrogen receptor status of the surgical specimen. A HR in the range of 1 to 2 receives one risk point; a HR in the 2 to 2.5 range, two risk points; a HR greater than 2.5, three risk points. The total risk point score for each patient is the sum of all the risk points accumulated from the four factors in the model, ranges from 0 (best possible outcome) to 12 (worst possible outcome).
Time Frame: At time of definitive surgery
Population: 2 participants in Group 1 did not have a PEPI score at time of surgery as (1) participant did not have nodal dissection and (1) did not have surgery. Both participants in Group 2 and Group 3 did not have surgery study tissue collected
Measure: Number; unit: participants
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Number analyzed (Participants) | 4 | 0 | 0
participants
  PEPI Score 1 | 1 |  |
  PEPI Score 4 | 1 |  |
  PEPI Score 7 | 1 |  |
  PEPI Score 8 | 1 |  |

5. Secondary Outcome: PEPI-0 Rate in Patients Whose Estradiol is Fully Suppressed (< or = 15 pg/mL) and Tumor Ki67 Level is 10% or Less
Time Frame: 16 weeks
Population: (1) of the participants in Group 1 had an inconclusive PEPI score at week 16 and was not evaluable. (1) of the participants in Group 1 did not have surgery and was not evaluable. Participants in Group 2 and Group 3 were not evaluable for this outcome as the estradiol and Ki67 levels were above outcome specified levels.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Number analyzed (Participants) | 4 | 0 | 0
percentage of participants | 0 |  |

ADVERSE EVENTS:
Arm/Group | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) | Group 3 (E2 > 15 pg/ml)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Ki67 <10%, E2 <= 15 pg/ml) (N=6) | Group 2 (Ki67 >= 10%, E2 <= 15 pg/ml) (N=1) | Group 3 (E2 > 15 pg/ml) (N=1)
Fatigue (General disorders) | 6 | 0 | 0
Chills (General disorders) | 3 | 0 | 0
Right heel pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hot flashes (Endocrine disorders) | 6 | 1 | 1
Night sweats (Endocrine disorders) | 5 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 0
Arthralgia (joint) (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 5 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Skin irritation around breast (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes